CLINICAL TRIAL: NCT05287659
Title: Low Calorie Diet or Very Low Calorie Ketogenic Diet Combined With Physical Training for Preserving Muscle Mass During Weight Loss in Sarcopenic Obesity
Brief Title: Low Calorie Diet or VLCKD Combined With Physical Training for Preserving Muscle Mass During Weight Loss in Sarcopenic Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Lucio Gnessi, Lucio Gnessi, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM2022SO
Record Dates: First submitted 2022-03-04; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenic Obesity
MeSH Terms: interventions — Dietary Supplements; Leucine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VLCKD group (Experimental): patients followed a structured VLCKD protocol (800Kcal/die)
  Interventions: Dietary Supplement: meal replacements or supplementation with leucine
- VLCKD and Physical Training group (Active Comparator): patients followed a structured VLCKD protocol (800Kcal/die) combined with interval training (IT), two times a week
  Interventions: Dietary Supplement: meal replacements or supplementation with leucine
- LCD and Leucine supplementation group (Active Comparator): patients followed a LCD regimen (1000 kcal/day) with supplementation of 18 g whey proteins which 4.1 g of leucine
  Interventions: Dietary Supplement: meal replacements or supplementation with leucine

INTERVENTIONS:
Dietary Supplement: meal replacements or supplementation with leucine — meal replacements or animal protein or supplementation with leucine

SUMMARY:
The prevalence of sarcopenic obesity (SO) is increasing worldwide, posing important challenges to public health and national health care system, especially during the COVID pandemic. In subjects with SO, it is essential to reduce body weight preserving lean mass, in order to avoid a worsening of muscle function. Lifestyle modification with adequate nutrition and proper physical activity is essential to counteract SO progression. In accordance with the Position Statement of the Italian Society of Endocrinology, Very Low Calorie Ketogenic Diet (VLCKD), a well established nutritional intervention in the context of obesity, has been promoted also for the treatment of SO. Moreover, the source of protein, timing of intake, and specific amino-acid constitution also represent critical factors in increasing muscle mass and strength. Recent studies have shown how protein supplementation, especially with high leucine content, can be effective in degenerative and end-stage diseases.

To date, the effects of physical training during VLCKD have not been studied. The aim is to determine the efficacy of VLCKD combined with interval training, compared to a VLCKD or a LCD alone, on weight-loss, body composition and physical performance in patient with SO.

ELIGIBILITY:
Inclusion Criteria:

* obesity (BMI 30-40)
* FAT MASS % ( > 41% for W, >29% for M)
* HOMA-IR > 2,5

Exclusion Criteria:

* known hypersensitivity to one or more components used in the protocol products; history of renal, cardiac or cerebrovascular diseases; psychiatric disturbances; hydroelectrolytic alterations, diagnosis of type 1 diabetes lack of informed consent; history of or planned weight loss surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Body weight | Body weight will be calculated at baseline and after 45 days
  Body weight change from baseline

SECONDARY OUTCOMES:
Body Mass Index | Body Mass Index will be calculated at baseline and after 45 days
  Body Mass Index change from baseline
Fat Mass | Fat Mass will be calculated at baseline and after 45 days
  Fat mass percentage (%) change from baseline
Fat Free Mass | Fat Free mass will be calculated at baseline and after 45 days
  Fat Free mass percentage (%) change from baseline
Fasting glucose | Fasting glucose will be calculated at baseline and after 45 days
  Fasting glucose level (mg/dL) change from baseline
Fasting insulin | Fasting insulin will be calculated at baseline and after 45 days
  Fasting Insulin level (mcU/mL) change from baseline
Muscle strength | Muscle strength will be calculated at baseline and after 45 days
  Muscle strength (kg) change from baseline
Physical Performance assessed by Short Physical Performance Battery (SPPB) | SPPB will be calculated at baseline and after 45 days
  Physical Performance change from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No